CLINICAL TRIAL: NCT05040750
Title: Correlation Between Cardiac Markers and Severity of COVID-19 in Egyptian Population
Brief Title: Correlation Between Cardiac Markers and Severity of COVID-19
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Maher Hussien, MD, Assistant professor of Anaesthesia, Ain Shams University
Other Study IDs: FMASU R 150 / 2021
Record Dates: First submitted 2021-09-09; First posted 2021-09-10 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Event
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- moderate to severe COVID 19 patients: moderate to severe COVID 19 patients admitted to ICU. Both genders within the age group 18-60 years were included. Diagnosis of COVID 19 was confirmed
  Interventions: Other: laboratory investigation

INTERVENTIONS:
Other: laboratory investigation — observe the relation between cardiac markers and mortality rate in critically ill COVID 19 patients

SUMMARY:
By July 9, 2020, the global pandemic of coronavirus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection had resulted in over 11.8 million confirmed cases and over 545000 deaths. Patients with a history of cardiovascular disease are especially vulnerable and have a bad prognosis. According to the findings, cardiac injury manifested by cardiac biomarker elevation is detected in a significant number of COVID-19 patients and is linked to poor outcomes and mortality. However, it is unclear how effective cardiac biomarkers are in COVID-19 prognosis and how to use these indicators.

DETAILED DESCRIPTION:
The pandemic of coronavirus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection has led to >11.8 million confirmed cases with >545000 deaths worldwide by July 9, 2020 Patients with preexisting cardiovascular conditions are particularly at risk and have poor prognosis data suggest that cardiac injury, manifested by cardiac biomarker elevation, is detected in a sizable of COVID-19 patients and is associated with adverse outcomes and increased mortality. However, how useful cardiac biomarkers are in COVID-19 prognosis and how to utilize these markers have not been well defined The study will include all moderate to severe COVID 19 patients admitted to ICU. Both genders within the age group 18-60 years were included. The primary outcome is the relation between cardiac markers and mortality rate in critically ill COVID 19 patients The secondary outcome is the relationship between cardiac and inflammatory and coagulation markers

ELIGIBILITY:
Inclusion Criteria:

* all moderate to severe COVID 19 patients who were admitted to ICU.
* Both genders
* age group 18-60 years

Exclusion Criteria:

* a refusal to participate in the study,
* pregnant patients,
* patients aged <18 or >60. years,
* recent history of acute myocardial infarction (< 1 month before admission).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: all moderate to severe COVID 19 patients who were admitted to ICU
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
relation between cardiac markers and mortality rate in critically ill COVID 19 patients | 4 month
  relate cardiac biomarkers to mortality rate

SECONDARY OUTCOMES:
relation ship between cardiac and inflammatory and coagulation markers | 4 month
  compare cardiac markers to inflammatory and coagulation laboratory findings

CONTACTS AND LOCATIONS:
Overall Officials: Fathy Tash, MD, Study Chair — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt